CLINICAL TRIAL: NCT03873311
Title: The Efficacy and Safety of Azacytidine Combined With HAG Regimen Versus Azacytidine for Elderly Patients With Newly Diagnosed Myeloid Malignancy: a Prospective, Randomized Controlled Trial
Brief Title: Azacytidine + HAG Regimen vs. Azacytidine for Elderly Patients With Newly Diagnosed Myeloid Malignancy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190109
Record Dates: First submitted 2019-03-08; First posted 2019-03-13 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukaemia; Myelodysplastic Syndromes;Chronic Myelomonocytic Leukemia
Keywords: Azacytidine; HAG regimen
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azacytidine + HAG Regimen (Experimental): Azacytidine（75mg/m2 ）+ HAG Regimen（Homoharringtonine(HHT) 1mg/(m2.d) , Cytarabine 10mg/(m2.d), G-CSF 200ug/(m2.d) )
  Interventions: Drug: Azacytidine, HAG Regimen
- Azacytidine (Active Comparator): 75mg/m2
  Interventions: Drug: Azacytidine

INTERVENTIONS:
Drug: Azacytidine, HAG Regimen — Azacytidine（75mg/m2 QD for 7 days）+ HAG Regimen（Homoharringtonine(HHT) 1mg/(m2.d) for 14 days), Cytarabine 10mg/(m2.d) for 14 days, granulocyte colony-stimulating factor(G-CSF) 200ug/(m2.d) for 14 days until absolute neutrophil count(ANC) ≥ 10X109／L)
  Other Names: Azacytidine, HAG Regimen (HHT Cytarabine G-CSF)
  Arms: Azacytidine + HAG Regimen
Drug: Azacytidine — Azacytidine 75mg/m2 QD for 7 days.
  Arms: Azacytidine

SUMMARY:
The primary objective is to explore the efficacy and safety of azacytidine and HAG regimen versus azacytidine for elderly patients with Newly Diagnosed MDS/AML/CMML in China. This is a post-marketing, interventional, multi-center, double-arm, prospective, open-label, randomized controlled study in elderly patients with MDS/AML/CMML in China. Patients will be recruited consecutively from the study sites during the enrollment period. The enrolled patients will be given azacytidine + HAG regimen or azacytidine under the conditions of informed consent and frequent monitoring according to the clinical guideline.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60;
* Patients with newly diagnoised diseases including MDS/AML/CMML;
* The ECOG behavior status score is less than 3 points;
* Agree to sign informed consent

Exclusion Criteria:

* Patients with a history of sever heart disease;
* Patients with severe organ dysfunction;
* Patients with other malignancies
* Patients who are allergic to the treatment of drug ingredients

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants (Responders) Achieving Overall Response Rate(ORR) After the Fourth Cycle Treatments. | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No